CLINICAL TRIAL: NCT00984841
Title: Can Tailored Patient Letters Improve The Quality Of Diabetic Patient Care?"
Brief Title: Can Tailored Patient Letters Improve The Quality Of Diabetic Patient Care?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scranton-Temple Residency Program (Other)
Responsible Party: John R Guzek, MD, Scranton-Temple Residency Program
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STRP001
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus targeted mailing
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored letter (Experimental): Patients in the tailored letter group received by mail a tailored letter detailing their diabetes measures, together with enclosed orders for lab tests when due, and reminder of or scheduling for an office appointment.
  Interventions: Other: Tailored letter
- Usual Care (Active Comparator): Patients in the usual care group were part of a practice wide quality improvement process.
  Interventions: Other: Tailored letter

INTERVENTIONS:
Other: Tailored letter

SUMMARY:
The purpose of this study is to determine if tailored letters sent to diabetic patients will improve care of diabetes.

DETAILED DESCRIPTION:
Diabetes care in the US is less than optimal. Some authors have found that targeted patient letters are also an effective tool to improve outcomes when they are part of a comprehensive disease management plan. Local patient satisfaction surveys had revealed that many patients had sub-optimal understanding of diabetes measures and of the importance of controlling these measures to reduce diabetic complications. We wondered if tailored patient letters and enclosed lab orders when due might increase patient awareness of diabetes measures and increase patient engagement.We hypothesized that the addition of targeted patient letters with enclosed lab orders to an ongoing performance improvement program would further improve diabetes care.

We conducted a randomized controlled study of tailored patient letters and diabetes lab orders at our two resident-based clinics.

ELIGIBILITY:
Inclusion Criteria:

* All active patients age 18 to 75 years with a diagnosis of diabetes mellitus were eligible.
* An active patient was defined as one having an ICD-9 code on the active problem list identifying the patient as diabetic, and a progress note in the EMR associated with an office visit within the prior 12 months.

Exclusion Criteria:

* None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Diabetes summary quality measure | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: John R Guzek, MD, Principal Investigator — Scranton-Temple Residency Program
Locations (1):
- Scranton-Temple Health Center, Scranton, Pennsylvania, United States